CLINICAL TRIAL: NCT04112862
Title: Effects of Sodium Lactate Infusion in Patients With Glucose Transporter 1 Deficiency Syndrome (GLUT1DS)
Brief Title: Sodium Lactate Infusion in GLUT1DS Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109147
Record Dates: First submitted 2019-09-18; First posted 2019-10-02 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-02

CONDITIONS: GLUT1 Deficiency Syndrome; GLUT1DS1; GLUT1DS2; Epilepsy; Lactic Acid Blood Increased; Ketogenic Dieting
Keywords: GLUT1 deficiency syndrome; sodium lactate infusion; epilepsy
MeSH Terms: conditions — Glut1 Deficiency Syndrome; Dystonia 18; Epilepsy; Hyperlactatemia

STUDY DESIGN:
Intervention Model Description: Single center, interventional, explorative, open label, proof of principle study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): three GLUT1DS patients with drug resistant epilepsy who tried the ketogenic diet without any benefits.
  Interventions: Other: sodiumlactate

INTERVENTIONS:
Other: sodiumlactate — intravenous sodiumlactate 600mmol/L

SUMMARY:
This study investigates the effect of lactate infusion on epileptic discharges on EEG and seizure frequency in glucose transporter 1 deficiency syndrome (GLUT1DS) patients.

DETAILED DESCRIPTION:
In glucose transporter 1 deficiency syndrome (GLUT1DS) cerebral glucose uptake from the systemic blood circulation is limited, because of deficient transport of glucose across the blood-brain barrier by the transporter protein (GLUT1). Classically patients present with developmental problems, movement disorders and severe epilepsy. There is no curative treatment for GLUT1DS, and anti-epileptic drugs usually have little to no effect. The ketogenic diet, providing ketones as an alternative energy substrate for the brain is an effective treatment option for the epilepsy and movement disorders in many GLUT1DS patients. Unfortunately, not in all GLUT1DS patients the ketogenic diet has a positive effect and other treatment options for these patients are very limited.

Traditionally, lactate is seen as a waste product of glycolysis during anaerobic conditions and a marker of ischemia. Interestingly, research has shown the beneficial side of lactate as an energy source for different organs. It seems that the brain can indeed use lactate as an alternative energy metabolite, besides glucose and ketones. The aim of this study is to investigate whether lactate can be an alternative energy metabolite in the GLUT1DS brain, and reduce epileptic discharges on EEG when intravenously administered in patients with GLUT1DS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GLUT1DS and known in our center.
* Baseline characteristics include a high frequency of clinical seizures and epileptic discharges on EEG.
* History of trying ketogenic diet with good compliance without beneficial effects.
* Age > 6 years.
* Informed consent.

Exclusion Criteria:

* Additional medical condition or illness that impairs the patient's ability to participate in the study (for example actual treatment of a malignancy, active infection, poorly controlled diabetes mellitus, hypertension, organ failure, clinically significant haematological or biochemical abnormalities).
* Elevated serum sodium (> 145 mmol/L).
* Participation in another interventional study at start of the study or during the study.
* Presence of known panic disorders or a history of panic attacks.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Number of changes in epileptic discharges on EEG during the infusion of lactate. | 1 day
  All subjects have frequent epileptic discharges on EEG. We want to objectify the change in epileptic discharges on EEG during and after the infusion of sodium lactate.

SECONDARY OUTCOMES:
Change in seizure frequency clinical visible by caregivers during and after infusion of sodium lactate. | 1 day
  All subjects have frequent seizures, we want to see if these clinically visible seizures reduce during or after infusion with sodium lactate.
Concentration of lactate in blood during and after sodium lactate infusion | 1 day
Concentration of glucose in blood during and after sodium lactate infusion | 1 day
Concentration of sodium in blood during and after sodium lactate infusion | 1 day
Concentration of potassium in blood during and after sodium lactate infusion | 1 day
Concentration of bicarbonate in blood during and after sodium lactate infusion | 1 day
Concentration of chloride in blood during and after sodium lactate infusion | 1 day
pH in blood during and after sodium lactate infusion | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We want to include three patients, who all are there own control. If one of their EEGs shows interesting changes during or after lactate infusion, we plan to describe that in our article.